CLINICAL TRIAL: NCT00129896
Title: Open-label Phase I-II Clinical Trial to Evaluate Treatment With Myocet/Taxotere/Herceptin as Primary Chemotherapy Treatment for HER2neu Positive Breast Cancer Patients
Brief Title: Neoadjuvant Chemotherapy With Myocet/Taxotere/Herceptin for HER2 Positive Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Cephalon (Industry); Sanofi (Industry); Hoffmann-La Roche (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 2003-03
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Her2neu positive breast cancer.; Neoadjuvant treatment.
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myocet+Taxotere+Herceptin (Experimental): Myocet 50 mg/m2; Taxotere 60 mg/m2; Herceptín 4 mg/Kg (first dose) and in the following cycles 2 mg/Kg
  Interventions: Drug: Myocet; Drug: Taxotere; Drug: Herceptin

INTERVENTIONS:
Drug: Myocet — Myocet®: 60-75 mg/m² ASC (vía IV) día 1 / c3s for 6 cycles
  Other Names: Lyposomal Doxorubicin
Drug: Taxotere — Taxotere® 70-75 mg/m² ASC (vía IV) día 1 / c3s for 6 cycles
  Other Names: Docetaxel
Drug: Herceptin — Herceptin® (4) 2 mg/kg (vía IV) Semanal for 6 cycles
  Other Names: Trastuzumab

SUMMARY:
This is an open-label study to assess the efficacy and tolerability of the combination Myocet®/Taxotere®/Herceptin® as primary treatment for HER2 positive breast cancer patients. HER2 status will be confirmed centrally by fluorescence in situ hybridization (FISH).

Phase I: Initial doses will be:

Myocet: 50-60 mg/m² day 1 every 3 weeks; Taxotere 60-75 mg/m² day 1 every 3 weeks; and Herceptin (4) 2 mg/kg weekly.

Sample size will depend on the number of patients recruited during dose escalation. Three patients must be recruited in each dose level. If one out of three experiences a dose-limiting toxicity (DLT), 3 more patients must be recruited in the same dose level. Considering that there are 4 dose levels to be tested, the estimated number of patients is 9 to 24. Patients receiving the recommended dose (RD) will be incorporated into phase II of the study.

DETAILED DESCRIPTION:
Phase II: The average pathological complete response rate reported in other trials is around 11%. The investigators expect to achieve an increase of 14% on this rate; that is, they expect a pathological response rate of 25%. With a= 0.05 and β=0.2, 18 patients are initially needed. If at least 3 pathological complete responses are achieved, recruitment will continue to up to 53 patients. At least 10 pathological complete responses are needed to probe the hypothesis. Considering a 10% post-randomization drop-out rate, a total of 59 patients must be recruited for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Breast cancer stages II and IIIA with histological diagnoses by true-cut.
* Breast cancer tumours overexpressing HER2neu, centrally confirmed by FISH.
* No evidence of metastasis: bilateral mammography, thorax x-ray, computed tomography (CT)-scan or abdominal echography and bone scintigraphy.
* Estrogen and progesterone hormone receptor status, determined before study registration.
* Age >= 18 years old.
* Performance status (Karnofsky index) >= 80.
* Adequate cardiac function by LVEF in the previous 14 days.
* Hematology: neutrophils >= 2.0 x10^9/l; platelets >= 100 x10^9/l; hemoglobin >= 10 g/dl.
* Adequate hepatic function: total bilirubin <= 1x upper normal limit (UNL); SGOT and SGPT <= 2.5xUNL; alkaline phosphatase <= 2.5xUNL.
* Adequate renal function: creatinine <= 1xUNL; creatinine clearance >= 60 ml/min.
* Patients able to comply with study treatment and follow-up.
* Negative pregnancy test in the previous 14 days.
* Adequate contraceptive method during the study and up to 3 months after definitive surgery.

Exclusion Criteria:

* HER2neu negative tumours.
* Prior systemic therapy for breast cancer.
* Prior treatment with anthracyclines or taxanes (paclitaxel, docetaxel) for any previous malignancy.
* Prior radiotherapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant or lactating women.
* Previous grade >= 2 motor or sensorial neurotoxicity (National Cancer Institute Common Toxicity Criteria [NCI CTC]).
* Other serious comorbidities: congestive heart failure or unstable angina; prior history of myocardial infarction in previous year; uncontrolled hypertension (HT); high risk arrhythmias; history of significant neurological or psychiatric disorders; uncontrolled active infection; active peptic ulcer; unstable diabetes mellitus; dyspnea at rest; or chronic therapy with oxygen.
* Previous or current history of neoplasms different from breast cancer, except for skin carcinoma, cervical in situ carcinoma, or any other tumor curatively treated and without recurrence in the last 10 years; ductal in situ carcinoma in the same breast; lobular in situ carcinoma.
* Chronic treatment with corticosteroids.
* Contraindications for administration of corticosteroids, anthracyclines, docetaxel, trastuzumab or egg derivates.
* Concomitant treatment with other therapy for cancer.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Tolerability (Phase I): Recommended Doses of the combination treatment | up to 24 months since last patient included in the Phase I
  Recommended Doses of the combination treatment
Efficacy (Phase II): Percentage (%) pathological Complete Response achieved according to Miller and Payne Criteria | up to 24 months since last patient included in the Phase II
  % pathological Complete Response achieved according to Miller and Payne Criteria

SECONDARY OUTCOMES:
Clinical response rates | up to 6 months since last patient treatment
  Clinical responses evaluated by radiological imaging
Surgery type (conservative surgery versus mastectomy) | up to 7 months since last patient treatment
  % conservative or mastectomy surgery
Potential cardiac toxicity | up to 12 months since last patient included
  Left ventricular ejection fraction [LVEF] by multiple-gated acquisition [MUGA])
Safety: Adverse Events evaluated according to NCI CTC v2.0 | 24 months since last patient included
  Adverse Events evaluated according to NCI CTC v2.0
Post-surgery node status | up to 7 months since last patient treatment
  according to Miller and Payne Criteria
Molecular changes in blood and tissue exams | 24 months
  Different biomarkers evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Univesitario Miguel Servet
Locations (16):
- Spain (16):
  - Hospital Universitario Virgen de los Lirios, Alcoy, Alicante
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Althaia-Xarxa Assistencial de Manresa, Manresa, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Onkologikoa, Donostia / San Sebastian, Guipúzcoa
  - Hospital de la Ribera, Alzira, Valencia
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Infanta Cristina, Badajoz
  - Hospital Clinic i Provincial, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Anton A, Ruiz A, Plazaola A, Calvo L, Segui MA, Santaballa A, Munoz M, Sanchez P, Miguel A, Carrasco E, Lao J, Camps J, Alfaro J, Antolin S, Camara MC. Phase II clinical trial of liposomal-encapsulated doxorubicin citrate and docetaxel, associated with trastuzumab, as neoadjuvant treatment in stages II and IIIA HER2-overexpressing breast cancer patients. GEICAM 2003-03 study. Ann Oncol. 2011 Jan;22(1):74-79. doi: 10.1093/annonc/mdq317. Epub 2010 Jul 5. PMID 20603435
- [Result] Anton A, Ruiz A, Segui MA, Calvo L, Munoz M, Lao J, Sancho F, Fernandez L. Phase I clinical trial of liposomal-encapsulated doxorubicin citrate and docetaxel, associated with trastuzumab, as neo-adjuvant treatment in stages II and IIIA, HER2-overexpressing breast cancer patients. GEICAM 2003-03 study. Ann Oncol. 2009 Mar;20(3):454-9. doi: 10.1093/annonc/mdn663. Epub 2008 Dec 11. PMID 19074216
- See also: Click here for more information about this study: GEICAM 2003-03 — http://www.geicam.org